CLINICAL TRIAL: NCT04074200
Title: PREPARE: A PRospective Evaluation of Pain After Inguinal Hernia REpair
Brief Title: Pain and Quality of Life After Inguinal Hernia Repair
Acronym: PREPARE
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-IHP-2018
Record Dates: First submitted 2019-08-22; First posted 2019-08-29 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Open Inguinal Hernia Repair: These subjects will undergo an inguinal hernia repair using an open surgical approach.
  Interventions: Procedure: Open Inguinal Hernia Repair
- Laparoscopic Inguinal Hernia Repair: These subjects will undergo an inguinal hernia repair using a laparoscopic surgical approach.
  Interventions: Procedure: Laparoscopic Inguinal Hernia Repair
- Robotic-assisted Inguinal Hernia Repair: These subjects will undergo an inguinal hernia repair using a robotic-assisted surgical approach.
  Interventions: Device: Robotic-Assisted Inguinal Hernia Repair

INTERVENTIONS:
Procedure: Open Inguinal Hernia Repair — With the patient under anesthesia, a single incision is made in the groin area. The hernia defect may be closed, as per the operating surgeon's standard of care (SOC). Mesh may be used to repair the hernia, as per SOC. The specific open approach may vary due to surgeon preference and patient characteristics. After the repair, the patient will be prescribed a 5 day supply of pain medication, as per SOC.
  Groups: Open Inguinal Hernia Repair
Procedure: Laparoscopic Inguinal Hernia Repair — With the patient under general anesthesia, several small incisions are made in the groin area. Ports are placed, the abdomen is insufflated, and laparoscopic instruments as well as a laparoscope (a lighted scope used to visualize the hernia) are inserted to complete the repair. The hernia defect may be closed, as per the operating surgeon's standard of care (SOC). Mesh may be used to repair the hernia, as per SOC. The specific laparoscopic approach may vary due to surgeon preference and patient characteristics. After the repair, the patient will be prescribed a 5 day supply of pain medication, as per SOC.
  Groups: Laparoscopic Inguinal Hernia Repair
Device: Robotic-Assisted Inguinal Hernia Repair — With the patient under general anesthesia, several small incisions are made in the groin area. Ports are placed, the abdomen is insufflated, and the da Vinci Robotic Surgical System (Intuitive) is docked to the patient and used to complete the procedure. The hernia defect may be closed, as per the operating surgeon's standard of care (SOC). Mesh may be used to repair the hernia, as per SOC. The specific robotic-assisted approach may vary due to surgeon preference and patient characteristics. After the repair, the patient will be prescribed a 5 day supply of pain medication, as per SOC.
  Groups: Robotic-assisted Inguinal Hernia Repair

SUMMARY:
This study aims to explore the difference in outcomes relating to pain and quality of life after open, laparoscopic, and robotic-assisted inguinal hernia repair.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational pilot study comparing outcomes of pain and quality of life after inguinal hernia repair between open, laparoscopic, and robotic-assisted surgical approaches. The study will focus on short-term outcomes through 3 months post-operation. During the post-operative period through 3 months, pain medication intake, pill count, subject-reported pain (on post-operative days 1-3 and 14 days post-surgery), and quality of life (at 14 days, 30 days, and 3 months post-surgery), incidence of intra- and post-operative complications, and time to return to normal activity will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 80 years of age.
* Subject is a candidate for an elective primary inguinal hernia repair.

Exclusion Criteria:

* Subject receiving a bilateral open repair.
* Subject who will have an emergent hernia repair.
* Subject with a history of chronic pain and/or taking daily pain medications for >6 weeks.
* Subject with a history of substance abuse and/or current (within 30 days) narcotic use.
* Subject with a history of methicillin-resistant Staphylococcus aureus (MRSA) infection.
* Diabetic subjects requiring insulin.
* Subject with recurrent hernias.
* Subject who will require the use of Exparel during the surgical procedure.
* Subject who will undergo a concomitant hernia repair or any other concomitant procedure.
* Current marijuana use that the subject is unwilling to discontinue within the 14 days prior to surgery.
* Subject is contraindicated for surgery.
* Subject has a known bleeding or clotting disorder.
* Pregnant or suspect pregnancy.
* Subject is mentally handicapped or has a psychological disorder or severe systemic illness that would preclude compliance with study requirements or ability to provide informed consent.
* Subject belonging to other vulnerable population, e.g, prisoner or ward of the state.
* Subject unable to comply with the follow-up visit schedule.
* Subject is currently participating in another research study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo an elective hernia repair procedure and meet all eligibility criteria will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scores from Baseline to 14 Days | 14 days post-surgery
  Change in patient-reported pain scores assessed by the Brief Pain Inventory Tool (BPI), with scores on individual questions ranging from 0% (no relief) to 100% (complete relief) or 0 (no pain/does not interfere) to 10 (pain as bad as you can imagine/completely interferes).
Change in Pain Scores from Baseline to 1 Day | 1 day post-surgery
  Change in patient-reported pain scores assessed by the Brief Pain Inventory Tool (BPI), with scores on individual questions ranging from 0% (no relief) to 100% (complete relief) or 0 (no pain/does not interfere) to 10 (pain as bad as you can imagine/completely interferes).
Change in Pain Scores from Baseline to 2 Days | 2 days post-surgery
  Change in patient-reported pain scores assessed by the Brief Pain Inventory Tool (BPI), with scores on individual questions ranging from 0% (no relief) to 100% (complete relief) or 0 (no pain/does not interfere) to 10 (pain as bad as you can imagine/completely interferes).
Change in Pain Scores from Baseline to 3 Days | 3 days post-surgery
  Change in patient-reported pain scores assessed by the Brief Pain Inventory Tool (BPI), with scores on individual questions ranging from 0% (no relief) to 100% (complete relief) or 0 (no pain/does not interfere) to 10 (pain as bad as you can imagine/completely interferes).
Change in Narcotic Usage from 1 Day Post-Surgery to 3 Months Post-Surgery | 3 months post-surgery
  Narcotic usage after the inguinal hernia repair procedure as determined by pill counts at study follow-up visits
Change in Narcotic Usage from 1 Day Post-Surgery to 30 Days Post-Surgery | 30 days post-surgery
  Narcotic usage after the inguinal hernia repair procedure as determined by pill counts at study follow-up visits
Change in Narcotic Usage from 1 Day Post-Surgery to 14 Days Post-Surgery | 14 days post-surgery
  Narcotic usage after the inguinal hernia repair procedure as determined by pill counts at study follow-up visits
Change in Narcotic Usage from 1 Day Post-Surgery to 7 Days Post-Surgery | 7 days post-surgery
  Narcotic usage after the inguinal hernia repair procedure as determined by patient Pain Diary completed at home

SECONDARY OUTCOMES:
Change in Over the Counter Pain Medication Usage from 1 Day Post-Surgery to 7 Days Post-Surgery | 7 days post-surgery
  Over the counter (OTC) pain medication usage after the inguinal hernia repair procedure as determined by patient Pain Diary completed at home
Change in Over the Counter Pain Medication Usage from 1 Day Post-Surgery to 3 Months Post-Surgery | 3 months post-surgery
  Over the counter (OTC) pain medication usage after the inguinal hernia repair procedure as determined by patient reporting of OTC pain medication usage at follow-up visits
Change in Over the Counter Pain Medication Usage from 1 Day Post-Surgery to 30 Days Post-Surgery | 30 Days post-surgery
  Over the counter (OTC) pain medication usage after the inguinal hernia repair procedure as determined by patient reporting of OTC pain medication usage at follow-up visits
Change in Over the Counter Pain Medication Usage from 1 Day Post-Surgery to 14 Days Post-Surgery | 14 Days post-surgery
  Over the counter (OTC) pain medication usage after the inguinal hernia repair procedure as determined by patient reporting of OTC pain medication usage at follow-up visits
Change in Quality of Life Assessment: EQ-5D-5L (EQ) from Baseline to 3 Months Post-Surgery | 3 months post-surgery
  Quality of life assessment using the EQ-5D-5L (EQ) assessment tool, with scores on individual questions ranging from no problems to extreme problems, with a scale of health ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Change in Quality of Life Assessment: EQ-5D-5L (EQ) from Baseline to 30 Days Post-Surgery | 30 Days post-surgery
  Quality of life assessment using the EQ-5D-5L (EQ) assessment tool, with scores on individual questions ranging from no problems to extreme problems, with a scale of health ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Change in Quality of Life Assessment: EQ-5D-5L (EQ) from Baseline to 14 Days Post-Surgery | 14 Days post-surgery
  Quality of life assessment using the EQ-5D-5L (EQ) assessment tool, with scores on individual questions ranging from no problems to extreme problems, with a scale of health ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Operative Time | Intra-operative
  Operative time, defined as first incision to closure of the incision
Length of Hospital Stay (LOS) | Admission to the hospital to discharge from the hospital (check out time), up to an approximate of one week
  How long the patient was admitted to the hospital
Conversion to Open | Intra-operative
  Incidence of conversions of the laparoscopic or robotic-assisted procedure
Number of Complications | Intra-operative through the 3 month follow-up period
  Intra-operative or post-operative complications related to the inguinal hernia repair

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No